CLINICAL TRIAL: NCT02110017
Title: Exploration of Neural Bases in Social Cognition
Acronym: IRM-COG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RCB 2013-A00064-41
Record Dates: First submitted 2013-09-12; First posted 2014-04-10 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Interpersonal Relations; Schizophrenia; Magnetic Resonance Imaging, Functional
Keywords: Ecological task; fMRI; Schizophrenia; Social Cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with schizophrenia (Other): Twenty patients suffering from schizophrenia (DSM-IV-R), with medication and medical care. No recent relapse of the psychotic disease, nor change in medications.
  No neurological comorbidity.
  After anatomic scans, each subject will go through the fMRI social cognition task.
  Interventions: Other: fMRI social cognition task
- Healthy subjects (Other): Twenty healthy subjects (no mental or neurological disease)
  After anatomic scans, each subject will go through the fMRI social cognition task.
  Interventions: Other: fMRI social cognition task

INTERVENTIONS:
Other: fMRI social cognition task — fMRI social cognition task : each subject will go through 3 runs of a fMRI paradigm, first one verbal then two visual runs, which are meant to activate the theory of mind network.
  Other Names: Philips 3 Tesla fMRI

SUMMARY:
An impairment in social cognition in schizophrenia could account for the severe professional and social difficulties among patients. Social cognition is the way the social world is understood, perceived and interpreted. It includes all the process than enable oneself to interact with another person, namely emotion perception and processing, theory of mind (ToM), social perception, social knowledge and attributional style. Since these process are interconnected, social cognition should be investigated through ecological tasks which activate all of them together. Developing a social cognition ecological task, then testing the reproducibility of the functional magnetic resonance imagery (fMRI) BOLD signal is the main objective of this study. The secondary objective is to seek a functional deficit among the neural network of social cognition in patients with schizophrenia compared with healthy subjects.

Forty healthy subjects, aged from 18 to 60 years old, who have given a written consent, will be included. The social cognition paradigm will be developed and the fMRI activations will be compared to those of a visual cartoon based task, known to turn on the neural network of ToM. BOLD signal variations at a high statistical correction ratio (p<0.05) will be explored and compared to the signal of a second fMRI, made on the same 20 healthy subjects one month later, to test reproducibility (% of identical activated voxels during the 2 fMRI, p<0.05).

Twenty matched patients with schizophrenia (DSM-IV-R), aged from 18 to 60 will be included to test the secondary objective. We make the hypothesis of a fMRI functional alteration in the cerebral network involved in social cognition, especially in the medial prefrontal cortex, among patients compared with healthy subjects.

DETAILED DESCRIPTION:
Social cognition neural basis. Impairment of the "social brain" in schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 18 to 60 years old
* who have signed a consent and, if there is one, whose legal representant has signed a consent

  1)For healthy subjects:
* without any psychiatric affection (Mini International Neuropsychiatric Interview)

  2)For patients
* meeting the DSM-IV-R criteria for schizophrenia or schizoaffective disorder

Exclusion Criteria:

* pregnant woman
* neurological affection
* medical objection to Magnetic Resonance Imagery (MRI)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Developing a social cognition ecological task, then testing the reproducibility of the functional magnetic resonance imagery (fMRI) BOLD signal | Day 1 for individual analysis. Up to 24 months for group analysis.
  The social cognition paradigm will be developed and the fMRI activations will be compared to those of a visual cartoon based task, known to turn on the neural network of ToM. BOLD signal variations at a high statistical correction ratio (p<0.05) will be explored and compared to the signal of a second fMRI, made on the same 20 healthy subjects one month later, to test reproducibility (% of identical activated voxels during the 2 fMRI, p<0.05)

SECONDARY OUTCOMES:
Identifying a functional deficit among the neural network of social cognition in patients with schizophrenia compared with healthy subjects. | Day 1 for individual analysis. Up to 24 months for group analysis.
  Using the previous social cognition ecological task, BOLD signal variations at a high statistical correction ratio (p<0.05) of 20 patients with schizophrenia will be compared to those of 20 matched healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Perrine BRAZO, MD-PhD, Principal Investigator — University of Caen, UMR 6301 ISTCT ISTS group; CNRS UMR 6301 ISTCT GIP Cyceron; CEA UMR 6301 ISTCT; CHU de Caen, Department of psychiatry, Centre Esquirol
Locations (1):
- Centre Hospitalier Universitaire, Caen, Normandy, France